CLINICAL TRIAL: NCT00625677
Title: A Phase IV, Randomized Study to Evaluate the Immune Response of UK Infants Receiving DTaP/Hib/IPV, Meningococcal C Conjugate and Pneumococcal Conjugate Vaccines, Antibody Persistence and Responses to Booster Doses in the Second Year of Life
Brief Title: Study to Evaluate the Immune Response of United Kingdom (UK) Infants Receiving DTaP/Hib/IPV, Meningococcal C Conjugate and Pneumococcal Conjugate Vaccines, Antibody Persistence and Responses to Booster Doses in the Second Year of Life
Acronym: Sched2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Public Health England (Other Government)
Collaborators: Institute of Child Health (Other); National Institute of Biological Standards and Control (Other Government)
Responsible Party: Prof Elizabeth Miller, Health Protection Agency
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Sched2; EudraCT No: 2007-004056-36
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2010-09

CONDITIONS: Meningococcal Infections; Pneumococcal Infections
Keywords: meningococcal serogroup C vaccine; reduced dose; meningococcal serogroup C conjugate vaccine; pneumococcal conjugate vaccine
MeSH Terms: conditions — Meningococcal Infections; Pneumococcal Infections | interventions — serogroup C meningococcal conjugate vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Pediacel - 2,3,4 months Prevenar - 2,4 months Menjugate - 3 months Hib/ pneumo conjugate/ Men C conjugate - 12 months
  Blood collected - 4,5,12,13 months
  Interventions: Biological: Menjugate (Meningococcal C conjugate vaccine)
- 2 (Experimental): Pediacel - 2,3,4 months Prevenar - 2,4 months Neis-vacC - 3 months Hib/ pneumo conjugate/ Men C conjugate - 12 months
  Blood collected - 4,5,12,13 months
  Interventions: Biological: NeisVacC (Meningococcal C conjugate vaccine)

INTERVENTIONS:
Biological: NeisVacC (Meningococcal C conjugate vaccine) — Dosage
  Other Names: Meningococcal C conjugate vaccine; Neis-vacC
  Arms: 2
Biological: Menjugate (Meningococcal C conjugate vaccine) — Dosage
  Other Names: Meningococcal C conjugate vaccine; Menjugate
  Arms: 1

SUMMARY:
The purpose of this study is:

To assess whether there are differences in antibody persistence eight months post primary (pre-booster) or in responses to the booster with regard to the Meningococcal C Conjugate (MCC) vaccine given in infancy.

To examine levels of diphtheria and tetanus antibody pre- and post-booster, with regard to the carrier proteins contained in the conjugate vaccines.

DETAILED DESCRIPTION:
There is a well recognised benefit in reducing the number of injections included in an immunisation programme, particularly for infants where delivery of many antigens in the first few months of life is essential in providing protection against deadly diseases. Reducing the number of injections would reduce distress to infants, parents and healthcare workers, make the schedule as cost effective as possible and would give greater flexibility to include vaccination against novel antigens in the future.

The UK recommended immunisation schedule up to 13 months of age was revised from 4 September 2006 so that infants receive three doses of Pediacel (diphtheria, tetanus, whooping cough, Hib and polio containing vaccine), two doses of Prevenar (pneumococcal vaccine, PNC) and two doses of meningococcal C vaccine, MCC, which can be one of three licensed products, Meningitec, Menjugate or NeisVacC. Previous studies have however shown that these three MCC products behave quite differently from each other when given with other vaccines and under different dose schedules. To that end the two products which seem viable as single dose options under the UK schedule, Menjugate and NeisvacC, will be included in this study.

Assessment of the absolute number of doses of vaccine needed to protect against disease essential in maximising the efficiency of the schedule and this study will further examine the dose requirement for meningococcal C conjugate (MCC) vaccine where there are data to suggest that this would be possible, both in the published peer reviewed literature and in an ongoing study conducted by our group. This study will be the first to test this under the accelerated UK schedule and in the presence of pneumococcal conjugate vaccine. This study also includes a booster phase where children receive a dose of MCC, PNC and Hib in the second year of life in accordance with the national schedule. There is a need for boosters in the second year of life to increase circulating antibody which has dropped significantly by a year of age. As expected, responses to boosting have been shown to be significantly higher than those achieved after primary immunisation with variation between products following a similar pattern to that seen with the primary series.

The current study is designed to allow assessment of a single dose of MCC vaccine given at three months of age for the two products that have shown potential to afford protection in the ongoing study above. In the previous study the first dose was given at two months of age and as responses tend to improve with age it is anticipated that this single dose being given later will result in higher antibodies than seen in the above study.

The aim of this study will be to provide data on which to base a decision about a further reduction in MCC vaccination in infancy from two doses to a single dose which would afford the benefits discussed above.

ELIGIBILITY:
Inclusion Criteria:

* No contraindications to vaccination as specified in the "Green Book" - Immunisation Against Infectious Disease, HMSO.
* Written informed consent obtained from the parent or legal guardian of the infant
* Infant aged no less than 7 weeks exactly, and no more than 11 weeks 6 days

Exclusion Criteria:

* None

Ages: 7 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 130 (Estimated)
Dates: Start 2008-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Miller, BSc MBBS FFPHM FRCPath, Principal Investigator — Public Health England
Locations (2):
- United Kingdom (2):
  - Health Protection Agency, Gloucester
  - Health Protection Agency, London

REFERENCES:
- [Result] Miller E, Andrews N, Waight P, Findlow H, Ashton L, England A, Stanford E, Matheson M, Southern J, Sheasby E, Goldblatt D, Borrow R. Safety and immunogenicity of coadministering a combined meningococcal serogroup C and Haemophilus influenzae type b conjugate vaccine with 7-valent pneumococcal conjugate vaccine and measles, mumps, and rubella vaccine at 12 months of age. Clin Vaccine Immunol. 2011 Mar;18(3):367-72. doi: 10.1128/CVI.00516-10. Epub 2010 Dec 29. PMID 21191076
- [Result] Borrow R, Andrews N, Findlow H, Waight P, Southern J, Crowley-Luke A, Stapley L, England A, Findlow J, Miller E. Kinetics of antibody persistence following administration of a combination meningococcal serogroup C and haemophilus influenzae type b conjugate vaccine in healthy infants in the United Kingdom primed with a monovalent meningococcal serogroup C vaccine. Clin Vaccine Immunol. 2010 Jan;17(1):154-9. doi: 10.1128/CVI.00384-09. Epub 2009 Nov 11. PMID 19906895
- [Result] Southern J, Borrow R, Andrews N, Morris R, Waight P, Hudson M, Balmer P, Findlow H, Findlow J, Miller E. Immunogenicity of a reduced schedule of meningococcal group C conjugate vaccine given concomitantly with the Prevenar and Pediacel vaccines in healthy infants in the United Kingdom. Clin Vaccine Immunol. 2009 Feb;16(2):194-9. doi: 10.1128/CVI.00420-08. Epub 2008 Dec 17. PMID 19091990